CLINICAL TRIAL: NCT00925405
Title: Breast MRI Screening in High-Risk Women After Mantle Radiation Therapy for Lymphoma
Brief Title: Breast Magnetic Resonance Imaging (MRI) Screening After Mantle Radiation Therapy
Status: Terminated | Type: Observational
Why Stopped: Low accrual
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Other Study IDs: 2009-0050
Record Dates: First submitted 2009-06-18; First posted 2009-06-22 (Estimated); Last update posted 2011-11-08 (Estimated); Status verified 2011-11

CONDITIONS: Breast Cancer
Keywords: Breast Cancer; Hodgkin's lymphoma; Mantle-field Irradiation; Mammogram; Magnetic resonance imaging; MRI Breast Cancer Screening
MeSH Terms: conditions — Breast Neoplasms; Hodgkin Disease

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Breast MRI Screening
  Interventions: Procedure: Breast MRI; Procedure: Mammogram

INTERVENTIONS:
Procedure: Breast MRI — Magnetic resonance imaging (MRI) scans of the breasts once per year
Procedure: Mammogram — Breast x-ray used to detect breast cancer and look for abnormalities in the breast.

SUMMARY:
Objectives:

The objective of this single-arm, prospective study is to perform annual mammography and MRI breast cancer screening in women who underwent mantle-field irradiation between 1970-1995 at M. D. Anderson Cancer Center in order to compare the ability of MRI and standard mammography to identify breast cancer. In addition, we will determine whether the combination of breast MRI and mammography identifies smaller, earlier-stage tumors, which would lead to improved cure rates. We will also take the opportunity to determine the incidence and stage of breast cancer in this high-risk cohort.

DETAILED DESCRIPTION:
Breast MRIs:

Breast MRIs have been reported to have higher sensitivity than mammograms for detecting early breast cancers, particularly in dense breasts where mammograms are not as effective. Although breast MRIs may add important information not provided by mammograms, the MRI must be used selectively. This is because the MRI is very sensitive and may show a false positive test (a test that shows cancer when there is none there).

Study Procedures:

If you are found to be eligible to take part in this study, the following procedures will be performed 1 time a year.

* You will have a breast exam.
* You will have a mammogram. A mammogram is a breast x-ray used to detect breast cancer and look for abnormalities in the breast.
* You will have an MRI of your breasts. For the MRI, you will lay on your stomach while a large donut-shaped scanner takes images of your breasts.

If any abnormality is found, you will have routine follow-up procedures performed. Routine follow-up may include additional imaging scans or biopsies. These will follow the standard of care, and the information will be collected and stored in your medical record.

Length of Study:

You will be on study for 20 years, with annual check-ups with breast imaging studies at M. D. Anderson. You will be taken off study if there is a change in your health that will not allow a breast mammogram or MRI, such as becoming pregnant.

This is an investigational study.

Up to 223 patients will take part in this study. All will be enrolled at M. D. Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Female patients diagnosed with lymphoma prior to 1995
2. The radiation therapy must have been delivered at M.D. Anderson from start to finish with complete records of dose received
3. Patients must have received radiation therapy to the chest between the ages of 10 and 30

Exclusion Criteria:

1. Patients with claustrophobia
2. Obese patients (the equipment weight limit is 350 pounds and the maximum scanner bore diameter is 55 cm)
3. Patients with myocardial infarction within 6 months of study entry
4. Patients with unstable angina pectoris, uncontrolled congestive heart failure, or uncontrolled arrhythmias
5. Patients with aneurysm clips, pacemakers, or other implanted devices that are not MRI compatible
6. Pregnant patients
7. Patients with compromised renal function, with a calculated glomerular filtration rate (cGFR) less than 60 ml/min/1.73m2.
8. Patients who began their treatment outside of MD Anderson Cancer Center.

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Women, breast cancer patients diagnosed with Hodgkin's lymphoma prior to 1995, who underwent mantle-field irradiation between 1970-1995 at M. D. Anderson Cancer Center.
Sampling Method: Non-Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2009-06; Primary Completion 2011-10 (Actual); Study Completion 2011-10 (Actual)

PRIMARY OUTCOMES:
Incidence of breast cancer detected with addition of breast MRI | Once a year

CONTACTS AND LOCATIONS:
Overall Officials: Bouthaina Dabaja, MD, Study Chair — UT MD Anderson Cancer Center
Locations (1):
- UT MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: UT MD Anderson Cancer Center website — http://www.mdanderson.org